CLINICAL TRIAL: NCT01415505
Title: A Multicenter, Open-Label, Single-Arm, Free Tablet Combination, Long-Term Study to Evaluate the Safety of Nebivolol in Combination With Valsartan in Patients With Stage 1 or Stage 2 Essential Hypertension
Brief Title: Combination of Nebivolol and Valsartan Given as Free Tablets for Stage 1 or Stage 2 Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAC-MD-02
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Hypertension
Keywords: Stage 1; Stage 2; Hypertension; 1 year open label safety study
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Valsartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Nebivolol and Valsartan free tablet combination
  Interventions: Drug: Nebivolol, Valsartan and Hydrochlorothiazide

INTERVENTIONS:
Drug: Nebivolol, Valsartan and Hydrochlorothiazide — Nebivolol 5 mg (tablet), oral administration Nebivolol 10 mg (tablet), oral administration Nebivolol 20 mg (tablet), oral administration Valsartan 160 mg (tablet), oral administration Valsartan 320 mg (tablet), oral administration Hydrochlorothiazide 12.5 mg rescue medication (capsules), oral administration. Hydrochlorothiazide 25 mg rescue medication (capsules), oral administration

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of nebivolol and valsartan given as a free tablet combination in patient with stage 1 or stage 2 essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients of age 18 years or above
* Patients diagnosed with stage 1 or stage 2 essential hypertension
* Normal physical examination findings, electrocardiogram (ECG) results and chest x-ray; or abnormal findings judged by the Investigator to be not clinically significant

Exclusion Criteria:

* Secondary hypertension or severe hypertension
* Clinically significant cardiovascular disease or heart failure
* A medical contraindication to discontinuing a current antihypertensive therapy
* History of Type 1 diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Adverse Event Recording | From Baseline to Week 53 (Visit 16)

SECONDARY OUTCOMES:
Diastolic Blood Pressure (DBP). | From Baseline to Week 52 (Visit 15)
Systolic Blood Pressure (SBP) | From Baseline to Week 52 (Visit 15)

CONTACTS AND LOCATIONS:
Overall Officials: David B Bharucha, MD, PhD, FACC, Study Director — Forest Laboratories
Locations (135):
- United States (135):
  - Forest Investigative Site 083, Birmingham, Alabama
  - Forest Investigative Site 004, Foley, Alabama
  - Forest Investigative Site 038, Gulf Shores, Alabama
  - Forest Investigative Site 124, Muscle Shoals, Alabama
  - Forest Investigative Site 023, Chandler, Arizona
  - Forest Investigative Site 073, Goodyear, Arizona
  - Forest Investigative Site 100, Green Valley, Arizona
  - Forest Investigative Site 117, Mesa, Arizona
  - Forest Investigative Site 065, Mesa, Arizona
  - Forest Investigative Site 102, Phoenix, Arizona
  - Forest Investigative Site 103, Tempe, Arizona
  - Forest Investigative Site 068, Tempe, Arizona
  - Forest Investigative Site 066, Jonesboro, Arkansas
  - Forest Investigative Site 118, Jonesboro, Arkansas
  - Forest Investigative Site 135, Carmichael, California
  - Forest Investigative Site 064, Encinitas, California
  - Forest Investigative Site 046, Encino, California
  - Forest Investigative Site 098, Glendale, California
  - Forest Investigative Site 129, Huntington Park, California
  - Forest Investigative Site 136, Lancaster, California
  - Forest Investigative Site 096, Long Beach, California
  - Forest Investigative Site 015, Los Angeles, California
  - Forest Investigative Site 025, Los Angeles, California
  - Forest Investigative Site 101, Mission Hills, California
  - Forest Investigative Site 089, Palm Springs, California
  - Forest Investigative Site 116, Pismo Beach, California
  - Forest Investigative Site 138, Sacramento, California
  - Forest Investigative Site 132, San Diego, California
  - Forest Investigative Site 061, San Marino, California
  - Forest Investigative Site 095, San Ramon, California
  - Forest Investigative Site 087, Santa Ana, California
  - Forest Investigative Site 134, Santa Barbara, California
  - Forest Investigative Site 062, Tustin, California
  - Forest Investigative Site 130, Tustin, California
  - Forest Investigative Site 092, West Hills, California
  - Forest Investigative Site 028, Westlake Village, California
  - Forest Investigative Site 006, Northglenn, Colorado
  - Forest Investigative Site 030, Cromwell, Connecticut
  - Forest Investigative Site 018, Waterbury, Connecticut
  - Forest Investigative Site 106, Boca Raton, Florida
  - Forest Investigative Site 044, Brooksville, Florida
  - Forest Investigative Site 049, Coral Gables, Florida
  - Forest Investigative Site 069, Cutler Bay, Florida
  - Forest Investigative Site 059, Daytona Beach, Florida
  - Forest Investigative Site 048, Fort Lauderdale, Florida
  - Forest Investigative Site 001, Fort Lauderdale, Florida
  - Forest Investigative Site 002, Hialeah, Florida
  - Forest Investigative Site 022, Miami, Florida
  - Forest Investigative Site 032, Miami, Florida
  - Forest Investigative Site 005, New Port Richey, Florida
  - Forest Investigative Site 021, North Miami Beach, Florida
  - Forest Investigative Site 111, Ocala, Florida
  - Forest Investigative Site 056, Pembroke Pines, Florida
  - Forest Investigative Site 127, Pembroke Pines, Florida
  - Forest Investigative Site 054, Pembroke Pines, Florida
  - Forest Investigative Site 133, Pembroke Pines, Florida
  - Forest Investigative Site 085, Plant City, Florida
  - Forest Investigative Site 033, Tampa, Florida
  - Forest Investigative Site 008, Winter Haven, Florida
  - Forest Investigative Site 019, Atlanta, Georgia
  - Forest Investigative Site 077, Roswell, Georgia
  - Forest Investigative Site 126, Arlington Heights, Illinois
  - Forest Investigative Site 084, Chicago, Illinois
  - Forest Investigative Site 088, Evansville, Indiana
  - Forest Investigative Site 108, Newton, Kansas
  - Forest Investigative Site 050, Lexington, Kentucky
  - Forest Investigative Site 003, Madisonville, Kentucky
  - Forest Investigative Site 141, Metairie, Louisiana
  - Forest Investigative Site 057, Auburn, Maine
  - Forest Investigative Site 041, Baltimore, Maryland
  - Forest Investigative Site 014, Baltimore, Maryland
  - Forest Investigative Site 080, Elkridge, Maryland
  - Forest Investigative Site 017, Haverhill, Massachusetts
  - Forest Investigative Site 143, Kalamazoo, Michigan
  - Forest Investigative Site 071, Troy, Michigan
  - Forest Investigative Site 086, Jackson, Mississippi
  - Forest Investigative Site 099, Omaha, Nebraska
  - Forest Investigative Site 120, Las Vegas, Nevada
  - Forest Investigative Site 119, Las Vegas, Nevada
  - Forest Investigative Site 121, Las Vegas, Nevada
  - Forest Investigative Site 137, Berkeley Heights, New Jersey
  - Forest Investigative Site 047, Binghamton, New York
  - Forest Investigative Site 072, Rosedale, New York
  - Forest Investigative Site 128, Saratoga Springs, New York
  - Forest Investigative Site 042, Charlotte, North Carolina
  - Forest Investigative Site 139, Greensboro, North Carolina
  - Forest Investigative Site 007, Hickory, North Carolina
  - Forest Investigative Site 114, Lenoir, North Carolina
  - Forest Investigative Site 081, Salisbury, North Carolina
  - Forest Investigative Site 013, Shelby, North Carolina
  - Forest Investigative Site 011, Wilmington, North Carolina
  - Forest Investigative Site 036, Winston-Salem, North Carolina
  - Forest Investigative Site 009, Cincinnati, Ohio
  - Forest Investigative Site 125, Kettering, Ohio
  - Forest Investigative Site 094, Marion, Ohio
  - Forest Investigative Site 093, Mount Gilead, Ohio
  - Forest Investigative Site 112, Oklahoma City, Oklahoma
  - Forest Investigative Site 104, Eugene, Oregon
  - Forest Investigative Site 058, Beaver, Pennsylvania
  - Forest Investigative Site 131, Penndel, Pennsylvania
  - Forest Investigative Site 105, Philadelphia, Pennsylvania
  - Forest Investigative Site 039, Upper Saint Clair, Pennsylvania
  - Forest Investigative Site 012, Charleston, South Carolina
  - Forest Investigative Site 040, Columbia, South Carolina
  - Forest Investigative Site 060, Greer, South Carolina
  - Forest Investigative Site 035, Mt. Pleasant, South Carolina
  - Forest Investigative Site 082, Mt. Pleasant, South Carolina
  - Forest Investigative Site 142, Simpsonville, South Carolina
  - Forest Investigative Site 045, Summerville, South Carolina
  - Forest Investigative Site 113, Bristol, Tennessee
  - Forest Investigative Site 034, Fayetteville, Tennessee
  - Forest Investigative Site 070, Franklin, Tennessee
  - Forest Investigative Site 016, Arlington, Texas
  - Forest Investigative Site 063, Carrollton, Texas
  - Forest Investigative Site 123, Dallas, Texas
  - Forest Investigative Site 079, Fort Worth, Texas
  - Forest Investigative Site 052, Houston, Texas
  - Forest Investigative Site 024, Houston, Texas
  - Forest Investigative Site 026, Houston, Texas
  - Forest Investigative Site 027, Houston, Texas
  - Forest Investigative Site 140, Plano, Texas
  - Forest Investigative Site 091, San Angelo, Texas
  - Forest Investigative Site 055, San Antonio, Texas
  - Forest Investigative Site 115, San Antonio, Texas
  - Forest Investigative Site 078, Sugar Land, Texas
  - Forest Investigative Site 090, Salt Lake City, Utah
  - Forest Investigative Site 053, Salt Lake City, Utah
  - Forest Investigative Site 051, St. George, Utah
  - Forest Investigative Site 110, Alexandria, Virginia
  - Forest Investigative Site 074, Burke, Virginia
  - Forest Investigative Site 067, Manassas, Virginia
  - Forest Investigative Site 037, Norfolk, Virginia
  - Forest Investigative Site 122, Suffolk, Virginia
  - Forest Investigative Site 010, Virginia Beach, Virginia
  - Forest Investigative Site 107, Tacoma, Washington

REFERENCES:
- [Derived] Neutel JM, Giles TD, Punzi H, Weiss RJ, Li H, Finck A. Long-term safety of nebivolol and valsartan combination therapy in patients with hypertension: an open-label, single-arm, multicenter study. J Am Soc Hypertens. 2014 Dec;8(12):915-20. doi: 10.1016/j.jash.2014.09.017. Epub 2014 Sep 28. PMID 25492835